CLINICAL TRIAL: NCT05618769
Title: Towards Life-Long Healthy Lungs: A Multidisciplinary Follow-up Framework for Preterm Infants (Dutch: Naar Levenslang Gezonde LONGen: Een multidiscipLinair zOrgpad Voor te Vroeg Geboren kindEren)
Brief Title: Towards Life-Long Healthy Lungs: A Multidisciplinary Follow-up Framework for Preterm Infants
Acronym: LONG LOVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Franciscus Gasthuis (Other)
Collaborators: Stichting BeterKeten (Unknown); Revenio Research (Industry); Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-117
Record Dates: First submitted 2022-10-03; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-09

CONDITIONS: Premature Birth; Respiratory Disease; Respiratory Tract Infections; Preterm Birth; Bronchopulmonary Dysplasia; Pollution Related Respiratory Disorder; Pollution; Exposure; Smoking Cessation; Health-Related Behavior; RSV Infection; RSV Pneumonia; Bronchial Hyperreactivity; Telemedicine; eHealth
Keywords: Moderate preterm; Late preterm; Post-Prematurity Respiratory Disease; Prematurity Associated Lung Disease; eHealth; mHeath; Follow-up; Respiratory Disease; Air pollution; Value Based Health Care
MeSH Terms: conditions — Premature Birth; Respiration Disorders; Respiratory Tract Infections; Bronchopulmonary Dysplasia; Smoking Cessation; Health Behavior; Respiratory Syncytial Virus Infections; Bronchial Hyperreactivity

STUDY DESIGN:
Intervention Model Description: Quasi-experimental design based on a non-randomized cluster trial, in which moderate-late preterm born infants will be allocated to the intervention or control group based on location of neonatal care. This design was chosen based on the limited amount of participating clusters and feasibility. As a quasi-experimental design can result in confounding by cluster and to increase internal validity, subjects of the control and intervention groups will be demographically matched at baseline
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (LONG LOVE Framework) (Experimental): Consists of participants born in Franciscus Gasthuis (FG) and/or Vlietland (FV) and will be allocated to the intervention group, receiving additional (in addition to current standard of care) follow-up in accordance with our newly developed framework to identify modi able influencing factors compromising pulmonary health using validated questionnaires, weekly monitoring of respiratory symptoms as reported by parents using an app, in- and outdoor air quality measurements and non-invasive pulmonary function measurements based on impedance pneumatography.
  In case of any modi able influencing factors, appropriate lifestyle and/or medical interventions will be undertaken.
  Interventions: Combination Product: LONG LOVE Framework
- Control (No Intervention): Consist of participants born in Maasstad Ziekenhuis (MSZ) and Albert Schweitzer Ziekenhuis (ASZ) and will receive standard of care follow-up.
  Parents are requested to provide informed consent for the registration of outcome measurements and requested to complete validated questionnaires. Data on utilization of medical services will be inquired to avoid recall bias.

INTERVENTIONS:
Combination Product: LONG LOVE Framework — In order to identify modifiable influencing factors, clinical data of the infants included in our multidisciplinary framework will be continuously collected by eHealth (Luscii Healthtech BV, Netherlands). Study visits take place at 1-1,5 3, 6, 12 and 18 months of age. Outdoor air quality measurements will be conducted using RIVM Luchtmeetnet. Indoor air quality measurements will be collected during a period of 6 weeks using a commercial available device. Lung function analysis using impedance pneumatography (Ventica Recorder, Revenio Research LTD, Finland) will take place during 2 nights at 3, 6 and 12 months of age. In the event of modifiable influencing factors medical or lifestyle interventions will be undertaken.
  Arms: Intervention (LONG LOVE Framework)

SUMMARY:
Approximately 8% of all births occur between 30-36 weeks of gestation ('moderate-late' prematurity). Respiratory tract infections (RTI) and wheezing illnesses disproportionally affect preterm infants resulting in a 1.5-2 fold higher hospitalisation rate during the first years of life compared to term born children. Besides prematurity, several other postnatal modifiable influencing factors are associated with increased risk of respiratory morbidity and impaired pulmonary development. These factors include RTI, rapid weight gain, air pollution, tobacco smoke exposition, vitamin D deficiency, maternal stress and antibiotic usage. The investigators hypothesize that a follow-up program aiming at prevention of modifiable influencing factors can reduce respiratory morbidity in moderate and late prematurity. Objectives: To reduce respiratory disease burden in moderate-late preterm infants in the first 18 months of life

DETAILED DESCRIPTION:
Background of the study:

Approximately 8% of all births occur between 30-36 weeks of gestation (moderate-late prematurity). Respiratory tract infections (RTI) and wheezing illnesses disproportionally affect preterms, resulting in a 1.5-2 fold higher hospitalization rate during the first years of life compared to term-born children. Besides prematurity, several other modifiable influencing factors are associated with increased risk of respiratory morbidity and impaired pulmonary development. These factors include rapid weight gain and obesity at an early age, tobacco smoke exposure, air pollution, microbiome composition, and recurrent RTI.

To promote optimal lung health and development in moderate-late preterm infants, increased respiratory health surveillance and protection against RTI in early life might be crucial. Previous research has shown that the introduction of a multidisciplinary follow-up framework in children with bronchopulmonary dysplasia resulted in a significant reduction in hospital readmissions.

Despite the burden of respiratory disease, moderate to late preterms do not currently receive standardised respiratory follow-up care. With LONG LOVE, the investigators introduce a novel follow-up framework tailored for preterms and designed to improve respiratory health. As the risk of the onset of pulmonary disease is further increased by postnatal factors such as tobacco smoke exposure, air pollution and RTI, our main focus is the detection and treatment of these modifiable influencing factors. LONG LOVE incorporates eHealth and new technology in order to measure pulmonary function and air quality. Intervention strategies include counseling on nutrition, lifestyle, medication, and improving indoor air quality.

Objective of the study:

The project's overarching aim is to diminish respiratory disease burden in moderate-late preterm born infants in their first 18 months of life.

The investigators have formulated the following specific objectives:

1. Determine whether the introduction of our follow-up framework will reduce the number and/or severity of RTI and wheezing episodes in the first 18 months of life
2. Analyse the predictive value of nocturnal impedance pneumatography on lower respiratory symptoms in prematurely born infants < 1 year of age. Further, correlate this novel tool to other forms of pulmonary function analyses such as the Lung Clearance Index and Hypoxic Challenge Test.
3. Conduct a cost-benefit analysis after the implementation of our framework.

Study design:

The investigators intend a quasi-experimental design based on a non-randomized cluster trial, in which moderate-late preterm-born infants will be allocated to the intervention or control group based on the location of birth. This design was chosen based on the limited amount of participating clusters and feasibility. As a quasi-experimental design can result in confounding by cluster and to increase internal validity, subjects of the control and intervention groups will be demographically matched at baseline[54,55]

Cluster 1 Consists of participants born in Franciscus Gasthuis (FG) and/or Vlietland (FV) and will be allocated to the intervention group, receiving additional (in addition to the current standard of care) follow-up in accordance with our newly developed framework to identify modifiable influencing factors compromising pulmonary health using validated questionnaires, weekly monitoring of respiratory symptoms as reported by parents using an app, in- and outdoor air quality measurements and non-invasive pulmonary function measurements based on impedance pneumatography.

In case of any modifiable influencing factors, appropriate lifestyle and/or medical interventions will be undertaken.

Cluster 2 (control) Consist of participants born in Maasstad Ziekenhuis (MSZ) and Albert Schweitzer Ziekenhuis (ASZ) and will receive standard of care follow-up.

Parents are requested to provide informed consent for the registration of outcome measurements and requested to complete validated questionnaires. Data on utilization of medical services will be inquired to avoid recall bias.

Study population:

Moderate-late preterm infants (GA 30+0-35+6 weeks) without other significant underlying syndromal, cardial, and/or pulmonal morbidities.

Intervention:

Follow-up regimen after premature birth using the LONG LOVE framework:

Identification of modifiable influencing factors Five study visits are scheduled to monitor health status on 1-1.5*, 3, 6, 12 and 18 months of age. These visits are planned in conjunction with regular follow-up examinations. Well-being and other potential risks will be determined by: growth, nutritional problems, feeding mode, pets, maternal stress (Edinburgh Postnatal Depression Scale questionnaire), sleep (Infant Sleep Questionnaire (ISQ)), tobacco smoke exposure, daycare attendance, the existence of siblings.

Air quality measurements Outdoor air analysis will be obtained using national and regional air measurement networks (RIVM Luchtmeetnet; DCMR Milieudienst Rijnmond). This network consists of a large number of air quality measurement sites, measuring harmful substances: nitric oxides (NOx, NO2), particulate matter (PM2.5, PM10), and ozone. Measurements will be taken from a station located nearest to the home address of the participant. Measurements are provided as publicly accessible data by the Dutch government.

Indoor air quality will be analyzed using a commercially available environment monitor. This device offers real-time monitoring of air quality factors such as temperature, humidity, particulate matter (PM1, PM2,5, PM10), carbon dioxide, and volatile organic compounds (VOCs). Air quality measurements will be taken from the living room or participants' sleeping room for a total duration of 1 year.

Pulmonary function analysis Pulmonary function analysis using impedance pneumatography will be measured at 3, 6, and 12 months of age during two consecutive nights using the Ventica recorder.

eHealth All parents are requested to install a newly developed application on their phones when enrolled in the study. The app is used for a weekly evaluation of respiratory symptoms. The following clinical parameters/variables will be monitored throughout the study: Respiratory health will be determined as follows: physician-diagnosed lower RTI- and wheezing episodes, hospitalizations for respiratory problems, clinical variables such as other respiratory episodes, common colds, medication use (bronchodilators, corticosteroids, antibiotics).

Interventions Aside from identification of potential health risks, our framework is designed to offer interventions if required. At baseline, all participants receive verbal and written information (App) defining potential hazardous factors regarding pulmonary development and overall health. In the event of pulmonary symptoms, parents are requested to consult a doctor.

In case of modifiable influencing factors, the following lifestyle and medical interventions will be performed:

In the case of 1.5 SDS weight gain or loss (based on birth weight), nutritional advice is provided by a paediatrician and follow-up by primary infant health care services.

In case of EPDS-scores ≥12 (stress-depression mother) consultation by lifestyle coach or community worker (Kleine Heldenhuis). If required, referral to general practitioner or psychologist/psychiatrist.

If sleep quality is affected (ISQ >12): medical advice and sleep training is provided by a paediatrician and/or primary infant health care services In the case of pulmonary symptoms: clinical assessment by a general practitioner or paediatrician. Administration of antibiotics according to Dutch board of Paediatricians guideline, optionally C-reactive protein measurement to prevent unnecessary antibiotics use If one or both caretakers are smoking: consultation by a general practitioner and primary infant health care services to provide stop-smoking services In case of inferior indoor air quality: visit by PhD-student or pulmonary care nurse to instruct how to improve air quality Optimal identification and treatment of comorbidity: gastro-oesophageal re ux disease, vitamin D deficiency, iron deficiency anaemia by paediatrician Active consultancy and treatment of nasal congestion using saline and-or xylometazoline by paediatrician Bronchodilator/broncholytic (salbutamol) trial by pediatrician in event of recurrent clinical bronchial obstruction and/or abnormal expiratory variability index using impedance pneumatography. If bronchodilator therapy is regularly required (a minimum of 2 episodes 2-3 days of week for a minimal duration of two weeks), inhaled corticosteroids can be prescribed.

These interventions are performed by both primary and secondary healthcare professionals (including the PhD-student who has an active role in patient management). Primary infant healthcare services operating in the Rijnmond region will fulfill an important role and are directly involved with the implementation of this framework.

ELIGIBILITY:
Inclusion Criteria:

* Moderate-late preterm infants (GA 30+0 - 35+6 weeks)

Exclusion Criteria:

* bronchopulmonary dysplasia (BPD)
* congenital diaphragmatic hernia (CHD),
* congenital pulmonary disorders
* hemodynamic significant cardiac disease
* immunodeficiency
* severe failure to thrive;
* birth asphyxia with poor neurological outcome
* syndromic or other severe congenital disorders with decreased life expectancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of lower Respiratory Tract Infections (RTI) | 18 months of life
  Total number of physician diagnosed lower RTI
Number of wheezing episodes | 18 months of life
  Total number of physician diagnosed wheezing episodes

SECONDARY OUTCOMES:
time to first lower RTI or wheezing episode | 18 months of life
  Elapsed time from birth until first RTI
total number of RTI | 18 months of life
  Total number of RTI
total number of wheezing episodes | 18 months of life
  total number of wheezing episodes
distribution of viruses (in case of hospital admission) | 18 months of life
  PCR measured viral distribution in case of hospital admission
medication use | 18 months of life
  Number of prescriptions (bronchodilators, corticosteroids, antibiotics)
lung function as measured by expiratory variability index (EVI) | 3, 6, 12 months of age
  Average EVI in preterm infants
comparison of expiratory variability index in moderate/late prematurity compared to term cohort (reference cohort from other center) | 3, 6, 12 months of age
  Average EVI
correlation between expiratory variability index and Lung Capacity Index and Hypoxic Challenge Test | 6 months of age
  EVI correlation with LCI and HCT
association between expiratory variability index and number of RTI/wheezing | 18 months of life
  association between low expiratory variability index and number of RTI/wheezing-rate
Analysis of outdoor air quality | 12 months
  Analysis of outdoor air quality using sensor and satellite data for increased spatial resolution: exceedance of health-based criteria (WHO, EU); outdoor-indoor pollution relationship; and association between air pollution and respiratory complaints/hospital admissions
indoor air quality | 12 months
  Analysis of indoor air quality using low-cost air quality sensors: exceedance of health-based criteria (WHO, EU), outdoor-indoor pollution relations; effect of direct feedback and strategies on optimization of indoor air quality
Preschool Children Quality of Life | 12 and 18 months of life
  by TNO-AZL Preschool Children Quality of Life (TAPQOL)
Total costs of framework | 18 months of life
  Total costs of framework consist of healthcare costs (medication and other healthcare costs), productivity costs and patient costs. Healthcare use will be assessed with the institute of Medical Technology Assessment (iMTA) Medical Consumption Questionnaire (iMCQ)supplemented with information on respiratory-related medication use, outpatient clinic visits and diagnostics extracted from the medical chart. Patient costs consisted of informal care and were measured using the iMTA MCQ. Healthcare and patient costs were valued according to the Dutch guideline. Productivity losses were estimated with the iMTA Productivity Cost Questionnaire (iPCQ)24 every 12 weeks. Productivity loss consists of absenteeism (sick leave), presenteeism (reduced effectiveness at work) and loss of unpaid work and will be evaluated using the iPCQ questionnaire
Care-related Quality of Life | 18 months of life
  Measuring and valuating the impact of providing informal care on caregivers using the CarerQoL questionnaire
Cost-effectiveness of framework | 18 months of life
  Societal costs as specified under 15 will be compared between both intervention and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Gerdien Tramper, MD, PhD, Principal Investigator — Franciscus Gasthuis & Vlietland
Locations (1):
- Franciscus Gasthuis & Vlietland, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided